CLINICAL TRIAL: NCT00201669
Title: A Phase II Study of Clofarabine in Patients With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0442
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Aggressive; Clofarabine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Aggression | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental)
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Clofarabine 30 mg/m2/day will be administered as a 2-hour intravenous infusion (IVI) on days 1-5.
  Other Names: Clolar

SUMMARY:
This study will determine the efficacy of clofarabine as measured by response rate in patients with aggressive non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
Rationale: Two Food and Drug Administration drugs approved for blood cancers such as non-Hodgkin's lymphoma (NHL) include fludarabine (Fludara) and cladribine (Leustat). The drug offered in the current study, clofarabine was designed to combine the anti-cancer strength of both fludarabine and cladribine. Laboratory research suggests that clofarabine targets anti-cancer mechanisms in cells, helps repair DNA, and inhibits tumor growth. Research also indicates that clofarabine has some efficacy against a variety of blood cancers and solid tumors. Numerous tumor responses have been observed with high doses of clofarabine in heavily pretreated patients with different types of lymphoma. The current study build on this previous research to test clofarabine in patients with aggressive NHL.

Purpose: This study will evaluate the safety and efficacy of clofarabine for aggressive NHL. Toxicities resulting from the combination of clofarabine and the supportive care drug GM-CSF will also be analyzed in patients. GM-CSF is a blood-forming agent that stimulates the production of white blood cells. In addition, several tests, including blood and tumor tissue analysis, will assess immune response and biological changes to the tumor as a result of study drugs.

Treatment: Patients in this study will be given clofarabine through intravenous infusions. This drug will initially be provided to patients for five consecutive days. Several tests will then be conducted and supportive care agents will be administered to stabilize patients' blood cell counts, immune response, and reduce the risk of infection. The first ten patients in this study will be hospitalized until recovery from the first five days of clofarabine to carefully monitor any additional toxicities resulting from the dosing regimen. Patients will receive another five day treatment cycle with clofarabine within seven days after recovering from each previous cycle and no more than four weeks from the start of the previous cycle. Disease response will be measured after every two cycles of treatment with clofarabine. Patient with stable or reduced disease will receive a maximum of six treatment cycles with clofarabine. Treatments will be discontinued due to disease growth, unacceptable side effects, or a treatment delay of more than 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed aggressive NHL
* B-cell NHL must be relapsed/ refractory
* T-cell & NK-cell and transformed lymphoma eligible at DX
* Patients with B-cell NHL (ie, diffuse large B-cell lymphoma, mantle cell lymphoma, and Burkitt's lymphoma) must have relapsed or refractory disease after at least 1 prior therapy.
* Patients previously treated with radioimmunotherapy (ie, ibritumomab tiuxetan [Zevalin] or tositumomab [Bexxar]) or prior stem cell transplant (SCT) are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Life expectancy of at least 12 weeks.
* Laboratory values obtained ≤ 7 days prior to registration:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelets ≥ 100,000/mm3
  * Total bilirubin ≤ upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 2 × ULN
  * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2 × ULN
  * Serum creatinine ≤ ULN

Exclusion Criteria:

* No prior treatment with clofarabine.
* Full recovery from all acute toxicities associated with prior chemotherapy, radiotherapy, or immunotherapy.- Patients with active, uncontrolled systemic infection considered to be opportunistic, life threatening, or clinically significant at the time of treatment or with a known or suspected fungal infection (ie, patients on parenteral antifungal therapy) are not eligible.
* Cardiac function (i.e. left ventricular ejection fraction) ≥ 50% on pretreatment radionuclide ventriculography (RVG) or echocardiogram.
* Women that are pregnant or breastfeeding.
* Known HIV disease.
* No CNS lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-10; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Response rate | up to two years

SECONDARY OUTCOMES:
Determine the toxicity of clofarabine administered in conjunction with growth factor support in patients with relapsed/refractory aggressive NHL. | up to two years
determine the effect of clofarabine on T-, B-, and natural killer (NK)-cell subsets and quantitative immunoglobulin levels after prolonged administration of clofarabine in patients with NHL. | up to two years
Assess cytokine (tumor necrosis factor [TNF]-alpha, interleukin [IL]-6, and IL-10) release following clofarabine therapy. | up to two years
Assess the effect of pre-treatment prognostic factors (p53 mutational status, DNA methylation, and apoptotic protein levels) in patient-derived tumor tissue on response to clofarabine. | up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu